CLINICAL TRIAL: NCT00762775
Title: The Interaction Between Calcium and Vitamin D Intake
Acronym: PTH Modified
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Winthrop University Hospital (Other)
Responsible Party: Principal Investigator, John F. Aloia, MD, Principal Investigator, Winthrop University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 33497; 08016
Record Dates: First submitted 2008-09-29; First posted 2008-09-30 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-12

CONDITIONS: Osteoporosis
Keywords: Bone resorption; Calcium homeostasis; Bone markers; Calcium and Vitamin D supplementation; Parathyroid hormone levels; Interaction between calcium and vitamin D supplementation
MeSH Terms: conditions — Osteoporosis; Bone Resorption | interventions — Calcium

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental): Calcium supplementation and placebo
  Interventions: Dietary Supplement: Calcium and vitamin D supplementation
- 2 (Experimental): Vitamin D supplementation and placebo
  Interventions: Dietary Supplement: Calcium and vitamin D supplementation
- 3 (Experimental): Calcium and Vitamin D supplementation
  Interventions: Dietary Supplement: Calcium and vitamin D supplementation
- 4 (Placebo Comparator): Placebos only
  Interventions: Dietary Supplement: Calcium and vitamin D supplementation

INTERVENTIONS:
Dietary Supplement: Calcium and vitamin D supplementation — Arm 1: 1,200 mg daily of calcium supplementation and placebo; Arm 2: 100 microgram daily of Vitamin D and placebo; Arm 3: 1,200 mg of calcium and 100 microgram of Vitamin D daily; Arm 4: placebos only.

SUMMARY:
We will study the relative importance of high calcium intake and vitamin D supplementation for calcium homeostasis, as determined by serum parathyroid hormone (PTH) and biochemical bone markers. We also intend to examine the interaction of vitamin D and calcium intake on calcium homeostasis. We hypothesize that optimal calcium supplementation and optimal vitamin D supplementation will lead to lower serum levels of PTH and markers of bone resorption compared with the placebo. We also theorize that when taken together, optimal calcium supplementation and optimal vitamin D intake will result in lower serum levels of PTH and bone markers compared with calcium or vitamin D taken alone.

ELIGIBILITY:
Inclusion Criteria:

* Healthy women aged 45 and above who have been menopausal at least 1 year (absence of menstrual period for a period of 12 months or more)

Exclusion Criteria:

* Any chronic medical illness including uncontrolled diabetes mellitus, recent history of myocardial infarction, or heart failure, malignancy, uncontrolled hypertension, obesity (BMI>35 kg/m2), history of anemia, leukemia, or other hematologic abnormalities, lupus, rheumatoid arthritis, or other rheumatologic disease, or kidney disease of any kind as determined by history and physical examination.
* Subjects with osteoporosis of the hip (total hip T-score equal or less than -2.5) or taking medications for osteoporosis such as bisphosphonates will be excluded.
* Pregnancy.
* Use of medication that influences bone metabolism (i.e. anticonvulsant medications, chronic use of steroids and high dose diuretics).
* Significant deviation from normal in medical history, physical examination, or laboratory tests as evaluated by the primary investigator.
* Patients with a history of hypercalciuria, hypercalcemia, nephrolithiasis, and active sarcoidosis will also be excluded.
* Participation in another investigational trial in the past 30 days prior to the screening evaluation.
* Unexplained weight loss of >15% during the previous year or history of anorexia nervosa.
* Medications that interfere with vitamin D metabolism.
* Patients with a habitual dietary calcium intake that exceeds 800 mg/day.
* Smokers greater than 1 pack per day will be excluded.
* Patients reporting alcohol intake greater than 2 drinks daily.
* Serum 25-hydroxyvitamin D level > 75 nmol/L.

Ages: 45 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2008-11; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
The influence of calcium supplementation alone on serum PTH levels and bone markers in healthy adult women. | 6 months

SECONDARY OUTCOMES:
The interaction between calcium and vitamin D supplementation and their combined effect on serum PTH hormone levels and bone markers in healthy adult women. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: John F. Aloia, MD, Principal Investigator — Winthrop University Hospital
Locations (1):
- Winthrop University Hospital, Mineola, New York, United States

REFERENCES:
- [Derived] Aloia JF, Dhaliwal R, Shieh A, Mikhail M, Islam S, Yeh JK. Calcium and vitamin d supplementation in postmenopausal women. J Clin Endocrinol Metab. 2013 Nov;98(11):E1702-9. doi: 10.1210/jc.2013-2121. Epub 2013 Sep 24. PMID 24064695